CLINICAL TRIAL: NCT07067398
Title: Improving the Cardiovascular Health of Home Health Aides
Brief Title: Improving the Heart Health of Home Health Aides
Acronym: VITAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 25-01028456; 23SCISA1142170 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2025-06-25; First posted 2025-07-16 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular; Cardiovascular (CV) Risk; Cardiovascular Disease (CVD) Risk Factors; Cardiovascular Health
Keywords: cardiovascular health intervention; home health aide; peer coaching
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Peer Coaching Delivered Life's Essential 8 Program (Experimental): Home Health Aides (HHAs) will receive educational content via paper-based booklets. HHAs will receive the 10-session adapted Life's Essential 8 program over 6 months. Each HHA will be paired with a trained Peer Coach participant who will work through the structured program with the HHA.
  Interventions: Behavioral: Peer Coaching Delivered Life's Essential 8 Program

INTERVENTIONS:
Behavioral: Peer Coaching Delivered Life's Essential 8 Program — This intervention includes structured bi-weekly peer coach (PC) Zoom or telephone sessions and a cardiovascular health curriculum including links to AHA resources. During the 1:1 session, PCs will elicit participants' challenges and successes from the previous week, track progress, and set goals (behavioral targets). PCs will use cognitive training techniques to teach participants how to manage negative thinking and replace it with positive thinking and goal setting. They will be encouraged to work towards these goals and monitor their progress (i.e. getting more physical activity on the job).

SUMMARY:
The goal of this early-stage study is to support the heart health of home health aides, a workforce that provides care for adults at home but whose own health has been historically poor. To do this, the study will use Life's Essential 8 (LE8), a program developed by the American Heart Association (AHA) that promotes cardiovascular wellness through education and lifestyle changes. The program has been adapted specifically for home health aides and will be delivered by trained "peer coaches," who are fellow home health aides who will help guide participants through the program.

The main questions the study aims to answer are:

* Will the LE8 intervention, which provides cardiovascular health education and support with positive thinking, be used by home health aides and do they like it?
* Does the LE8 intervention actually improve home health aides' cardiovascular health after the intervention's conclusion compared to baseline?

Participants will be paired with a trained peer coach and take part in the 10-week program over the course of 6 months. The program includes support for healthy behaviors and positive thinking, with the goal of making lasting improvements in cardiovascular health.

DETAILED DESCRIPTION:
The goal of the proposed project is to improve the cardiovascular (CV) health of home health aides and attendants (HHAs), one of the fastest growing sectors of the healthcare industry, comprised predominantly of middle-aged women of color with a high burden of CV disease risk factors, including obesity, hypertension, hyperlipidemia, physical inactivity, and smoking. Improving HHAs' cardiovascular health and well-being is not only critical to their own longevity as a workforce, but it has the potential to improve the health of the patients for whom they care. The overall goal of the study is to test the preliminary effectiveness of the peer-coach (PC) delivered Life's Essential 8 (LE8) intervention program among 40 HHAs with poor CV health, while gathering data on its implementation.

The investigators have 3 main hypotheses. Under Aim 1, the investigators hypothesize that HHAs who receive the intervention will have higher CV health at follow-up compared to baseline. Under Aim 2, the investigators hypothesize that drivers of implementation will include: intervention adaptability, local conditions, work infrastructure, recipient centeredness, and motivation. Also under Aim 2, the investigators hypothesize the intervention will be feasible (>80% HHAs complete the study) and acceptable (>90% HHAs high levels of satisfaction).

All aspects of the study, including the intervention itself, will be conducted using a hybrid (in-person and virtual) model, with some sessions being completed online and others in person. .

ELIGIBILITY:
Inclusion Criteria:

* Currently working as a home health aide
* Speak English or Spanish
* ≥ 18 years of age
* Have low CV Health as assessed by LE8 components made up by physical health measurements (blood pressure, BMI) and general self-reported health (physical activity, diet, smoking, sleep); calculated to be a score of 0-50 (the total score ranges from 0-100)

Exclusion Criteria:

* Less than 1 year of job experience as a home health aide
* Does not possess a smartphone
* Gotten dizzy before with a finger stick blood sugar/cholesterol test
* Have a history of syncope with a finger stick blood sugar/cholesterol test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Effectiveness, which will be assessed by a change from baseline in overall cardiovascular health score as measured by LE8. | From baseline to end of the intervention at 6 months
  Each individual Life's Essential 8 (LE8) domain (physical activity level, diet, smoking, sleep, and physiologic health (systolic and diastolic blood pressure), BMI, hemoglobin A1C, and non-HDL cholesterol) has a score of 0 to 100, with higher values indicating better cardiovascular health in each domain. The LE8 overall score is created by averaging individual scores across 8 domains. The overall score ranges from 0 to 100 with higher numerical values corresponding to better cardiovascular health.

SECONDARY OUTCOMES:
Implementation, which will be assessed by acceptability through a qualitative interview | One 30-90 minute session following the end of the intervention at 6 months
  Acceptability defined as participant satisfaction of the study will be assessed through a qualitative interview
Implementation, which will be assessed by acceptability through a survey | Following the end of the intervention at 6 months
  Acceptability will be assessed through the 4-item, validated, Acceptability of Intervention Measure. Items are measured on a 5-point Likert scale (Completely Disagree-Completely Agree). The score is calculated as the mean. The scale for this measure ranges from 4-20 with higher scores indicating greater perceived acceptability of the intervention.
Implementation, which will be assessed by feasibility through a qualitative interview | One 30-90 minute session following the end of the intervention at 6 months
  We will ask peer coaches about the intervention's feasibility, or how viable it was considering their experience, through qualitative interviews.
Implementation, which will be assessed by feasibility through a process measure | Following the end of the intervention at 6 months
  Feasibility will be assessed with the number of HHAs eligible to receive the intervention.
Implementation, which will be assessed by feasibility through a process measure | Following the end of the intervention at 6 months
  Feasibility will be assessed with the number of HHAs who receive the intervention.
Implementation, which will be assessed by feasibility through a process measure | Following the end of the intervention at 6 months
  Feasibility will be assessed with the number of HHAs who completed the intervention.
Implementation, which will be assessed by feasibility through a process measure | Following the end of the intervention at 6 months
  Feasibility will be assessed with the number of additional staff needed for implementation determined as the study progresses.
Implementation, which will be assessed by feasibility through a survey | Following the end of the intervention at 6 months
  Feasibility will be assessed with a validated, 4-item, Feasibility of Intervention Measure. Items are measured on a 5-point Likert scale (Completely Disagree-Completely Agree). The score is calculated as the mean. The scale for this measure ranges from 4-20 with higher scores indicating greater perceived feasibility of the intervention.
Implementation, which will be assessed by fidelity through a process measure | From baseline to end of the intervention at 6 months
  Fidelity defined as number of subjects who adhered to the intervention as assessed with checklists tracking participants' completion of scheduled educational lessons.
Implementation, which will in part be assessed by adaptation through a process measure | From baseline to end of the intervention at 6 months
  Adaptation defined as number of changes made to the intervention during the study will be assessed by documenting how the intervention was modified and refined.
Effectiveness, which will be assessed by a change from baseline in well-being (quality of life) as measured by a survey | From baseline to end of the intervention at 6 months
  Social support will be assessed with a validated 4-items measure of perceived adequacy of social support from people in one's life and on the job. Items are measured on a 5-point Likert scale (Not at all-Very much). The score is calculated as the mean across items reported per day. Higher scores indicate greater perceived social support from colleagues and supervisors in response to daily work stressors.
Effectiveness, which will be assessed by a change from baseline in well-being (quality of life) as measured by a survey | From baseline to end of the intervention at 6 months
  Self-efficacy will be assessed with a validated, 10-item measure of one's confidence in handling situations related to health, job, personal life. Items are measured on a 4-point Likert scale (Not at all true-Exactly true). The score is calculated as the sum or mean of all items. The scale ranges from 10-40 (sum) or 1-4 (mean), with higher scores indicating greater perceived general self-efficacy.
Effectiveness, which will be assessed by a change from baseline in employment-related outcomes as measured by a survey | From baseline to end of the intervention at 6 months
  Job satisfaction will be assessed with a validated, 5-item measure that assesses satisfaction with current job. Items are measured on a 7-point Likert scale (Strongly Disagree-Strongly Agree). The score is calculated as the mean of all items. The scale ranges from 1-7, with higher scores indicating greater satisfaction with one's work.
Effectiveness, which will be assessed by a change from baseline in employment-related outcomes as measured by a survey | From baseline to end of the intervention at 6 months
  Turnover intention as an employment-related outcome will be assessed with a validated, 2-item measure that assesses likelihood to leave job. Items are measured on a 5-point Likert scale (Strongly Disagree-Strongly Agree). The score is calculated as the mean of all items. The scale ranges from 1-5, with higher scores indicating a stronger intention to leave one's job or the workforce.

CONTACTS AND LOCATIONS:
Overall Officials: Madeline Sterling, MD, MPH, MS, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - 1199 SEIU Home Care Industry Education Fund, New York, New York
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No